CLINICAL TRIAL: NCT02001129
Title: Improving Follow-Up Adherence in a Primary Eye Care Setting: A Prospective, Randomized Controlled Trial
Brief Title: Improving Follow-Up Adherence in a Primary Eye Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Julia Haller, Ophthalmologist-in-Chief, Wills Eye
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: WEF 14-040
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Eye Diseases
Keywords: Eye care adherence; health care utilization
MeSH Terms: conditions — Eye Diseases; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Automated Telephone System (Experimental): In addition to a standardized reminder letter, participants also received a telephone call from an automated system to remind them of a recommended follow-up appointment.
  Interventions: Behavioral: Personalized Telephone Call; Behavioral: Usual Care
- Personalized Telephone Call (Experimental): In addition to the usual care letter, a staff member called participants one month prior of recommended follow-up appointment. During this call, participants were given the option to schedule an appointment.
  Interventions: Behavioral: Automated Telephone System; Behavioral: Usual Care
- Usual Care (Active Comparator): Participants randomized to this arm receive a "usual care" letter which is a standard reminder letter from the primary eye care office. This is usual practice in many primary eye care facilities.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Automated Telephone System — Participants receive automated reminder phone calls.
  Other Names: Patient appointment message 2000
  Arms: Personalized Telephone Call
Behavioral: Personalized Telephone Call — Participants receive reminder phone calls by study staff.
  Other Names: Study staff phone call
  Arms: Automated Telephone System
Behavioral: Usual Care — Participants receive a standard reminder letter in the mail.
  Other Names: Reminder letter sent in the mail.

SUMMARY:
This study aims to examine the effectiveness of three different ways of helping patients attend their recommended eye care appointments.

DETAILED DESCRIPTION:
The three ways are 1) usual care, which involves a standard reminder letter; 2) automated telephone calls, which utilizes a machine to automatically call patients one month prior to their recommended follow-up date; 3)personalized telephone calls, which utilizes a staff member to personally call patients and offer them the opportunity to schedule at the time of the telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18 years
* Primary Eye Care Patients who were recommended for a 6-month, 12-month, or 24-month follow-up appointment during September 2013 through November 2013.
* Access to a telephone

Exclusion Criteria:

* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Appointment Adherence | 3 months
  A research assistant examines the Electronic Medical Records (EMR) system to assess recommended appointment adherence.

SECONDARY OUTCOMES:
Scheduling Appointment | 1 month
  Tracking whether the patient made an appointment within 1 month of the reminder letter (usual care), automated phone call, or personalized phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hark, PhD, Study Director — Wills Eye
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callinan CE, Kenney B, Hark LA, Murchison AP, Dai Y, Leiby BE, Mayro EL, Bilson J, Haller JA. Improving Follow-Up Adherence in a Primary Eye Care Setting. Am J Med Qual. 2017 Jan/Feb;32(1):73-79. doi: 10.1177/1062860615616860. Epub 2016 Jul 10. PMID 26656245